CLINICAL TRIAL: NCT06624761
Title: Determination of the Effect of Shotblocker in Reducing Intramuscular Injection Pain in Adult Patients: A Randomized Controlled Trial
Brief Title: Effect of Shotblocker in Reducing Intramuscular Injection Pain in Adult Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yağmur SÜRMELİ (Other)
Collaborators: Toros University (Other)
Responsible Party: Sponsor-Investigator, Yağmur SÜRMELİ, LECTURER DR., Mersin University
Organization: Mersin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-79438647-108-48697 TU
Record Dates: First submitted 2024-09-24; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Patients Above 18 Years
Keywords: ShotBlocker; intramuscular injection pain; nursing

STUDY DESIGN:
Intervention Model Description: There will be 2 groups (ShotBlocker and control )
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ShotBlocker (Experimental): ShotBlocker will be applied to the experimental group.
  Interventions: Device: ShotBlocker
- Control group (No Intervention): no intervention will be made

INTERVENTIONS:
Device: ShotBlocker — A randomized study investigating ShotBlocker in painkillers containing different active ingredients could not be found.
  Arms: ShotBlocker

SUMMARY:
This randomized, double-blind study aimed to determine the effect of ShotBlocker on IMI pain in adult patients who received diclofenac sodium and metamizole sodium as IMI in the emergency department. The main question(s) it aims to answer are as follows:

• [Is there a difference between the pain score averages between the intervention group and the control group after ShotBlocker? Participants [Participants in both groups are individuals who applied to the emergency department and received IM injections according to the doctor's order.] If there is a comparison group: Researchers will make a comparison with the control group.

DETAILED DESCRIPTION:
The study is planned to be conducted between October 2024 and December 2024. The population of the study will consist of adult patients who have applied to the emergency department of a state hospital in Turkey between October 2024 and December 2024 due to the use of previously prescribed drugs (diclofenac sodium and metamizole sodium) or who need to be administered IMI diclofenac sodium and metamizole sodium upon the order of the emergency room physician. The minimum sample size expected to complete the data collection form of the study was calculated with G power analysis at a 95% confidence level before the data collection phase. Accordingly, the sample size required for the study was determined as 25 for each group, with an alpha value of 0.01, an effect size of 1.583, and a theoretical power of 99% [23]. In case of sample loss during the study, it was planned to take 20% more samples than the calculated sample and to include 30 people in each group (with and without ShotBlocker).

As data collection tools; Personal and Applied Drug Information Form and Visual Analog Scale will be used. Personal Information Form will consist of 8 questions in total, 7 of which include the patients' introductory characteristics (age, gender, height, weight, fear of injection) and 1 question including the name of the drug. In addition to this form, Visual Analog Scale (VAS) is used to measure the pain perceived by the person. In this scale, the person can indicate his/her own pain by drawing a line, putting a dot or pointing between the part where there is no pain (zero) on one end of the ruler and the part where there is the most severe pain (10 cm) on the other end. The distance from the point where there is no pain to the point marked by the person is measured in centimeters and the value found indicates the person's pain intensity. In the VAS scale, 0-44 mm reflects mild pain, 45-74 mm reflects moderate pain and 75-100 mm reflects severe pain.

Research Application Procedure Step 1: Before starting the application, a preliminary interview will be conducted with practitioners who are not included in the study and who work as nurses in the emergency department. Information will be provided about the purpose of the study and the scale to be used. It will also be stated that these forms will be filled out by patients who received diclofenac sodium and metamizole sodium as IMI from the ventrogluteal region, used ShotBlocker during this period and met the research criteria.

Step 2: VAS will be applied to the patients immediately after the application. Step 3: VAS will also be applied to patients in the control group who received diclofenac sodium and metamizole sodium as IMI from the ventrogluteal region, did not use ShotBlocker during this period and met the research criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over who speak Turkish,
* Who have signed the informed consent form,
* Who are admitted to the emergency room for prescription drug use or who are planned to use diclofenac sodium and metamizole sodium as IMI upon the directive of the emergency room physician will constitute.

Exclusion Criteria:

* Pregnant women,
* Those with psychiatric disorders,
* Those with hearing or vision problems,
* Those who applied to the red area of the emergency room,
* Those with impaired consciousness,
* Those with secondary injuries and infections at the injection site,
* Those who have previously received an injection at the same site within the last 24 hours, -Those who did not sign the informed consent form for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-14 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 12 week.
  The Visual Analog Scale (VAS) is used to measure the pain perceived by the person. In this scale, the individual can indicate their own pain by drawing a line, putting a dot, or pointing between the 10 cm (100 mm) section of the ruler where there is no pain (zero) on one end and the most severe pain on the other end. The distance from the point where there is no pain to the point marked by the individual is measured in centimeters and the value found indicates the individual's pain intensity. On the VAS scale, 0-44 mm indicates mild pain, 45-74 mm indicates moderate pain, and 75-100 mm reflects severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: YAGMUR SÜRMELI, DR., Study Director — Toros University
Locations (1):
- Toros State Hospital, Mersin, Adana, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No